CLINICAL TRIAL: NCT04587518
Title: Five Factor Model Treatment for Borderline Personality Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shannon E. Sauer-Zavala (Other)
Responsible Party: Sponsor-Investigator, Shannon E. Sauer-Zavala, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 60042
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Borderline Personality Disorder
Keywords: borderline personality disorder; treatment; CBT; five-factor model
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate Treatment (Experimental): Participants in this group will receive the intervention immediately.
  Interventions: Behavioral: Personality-Based Cognitive Behavioral Therapy
- Waitlist/Delayed Treatment (Experimental): Participants in this group will receive the intervention after an 18-week wait.
  Interventions: Behavioral: Personality-Based Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Personality-Based Cognitive Behavioral Therapy — The study treatment will take place across 18-sessions. The first session will involve psychoeducation regarding BPD.The next two sessions with include exercises drawn from Behavioral Activation (i.e., identification of value-based goals) and Motivational Interviewing (i.e., pros and cons [long and short-term consequences] of tolerating emotions, engaging in prosocial behavior, and delaying gratification). Next, patients will receive 5 sessions of cognitive interventions (i.e., cognitive reappraisal related to situations/emotions, schema related to relationships, 5 sessions of behavior change skills (i.e., acting opposite to emotion-driven urges, exposure, assertiveness training), and 5 sessions of mindfulness skills (i.e., nonjudgmental emotion awareness, compassion training, urge surfing). Finally, treatment will conclude with 2 sessions of Relapse Prevention strategies. All sessions will last for 60 minutes in duration.

SUMMARY:
The primary purpose of this study is to explore acceptability, feasibility, and preliminary efficacy of a novel cognitive-behavioral treatment for borderline personality disorder (BPD). Extant treatments for this condition are intensive, long-term (usually at least one year), and have, understandably, focused on targeting the life-threatening and therapy-interrupting behaviors that often characterize this disorder. BPD, however, is a heterogeneous disorder with diagnostic criteria that can be combined to create over 300 unique symptom presentations (Ellis, Abrams, & Abrams, 2008); to date, no treatments have been explicitly designed with lower risk presentations of BPD in mind. This is unfortunate, as there is evidence to suggest that the majority of individuals with BPD do not demonstrate the recurrent life-threatening behaviors that warrant intensive, long-term care (Trull, Useda, Conforti, & Doan, 1997; Zimmerman & Coryell, 1989). Additionally, various studies have shown that the difficulties experienced by individuals with BPD can be understood as manifestations of maladaptive variants of personality traits (e.g., Mullins-Sweatt et al., 2012). Specifically, individuals with BPD demonstrate high levels of neuroticism, and low levels of agreeableness (antagonism) and conscientiousness (disinhibition); these traits may not be universally present across all individuals with BPD, perhaps underscoring the heterogeneity in presentations of this condition.

ELIGIBILITY:
Inclusion Criteria:

-diagnosis of borderline personality disorder (BPD)

Exclusion Criteria:

* diagnosed psychological conditions that would be better addressed by alternative treatments
* previously received more than 5 sessions of cognitive behavioral therapy in the past 5 years
* concurrent psychotherapy
* medication instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-03 (Actual)

PRIMARY OUTCOMES:
Change in clinician-rated borderline personality disorder symptoms | 44 weeks (baseline, post-treatment/waitlist, 6 month follow-up)
  Change in borderline personality disorder symptoms will be measured using Zanarini Rating Scale for Borderline Personality Disorder (ZAN-BPD) - clinician-rated version. Scores range from 0-36; higher scores indicate greater severity of borderline personality disorder symptoms
Change in patient-reported borderline personality disorder symptoms | 18 weeks (week 1[baseline for immediate treatment condition, post-waitlist for delayed treatment condition], week, 2, week 3, week, 4.....week 18)
  Change in borderline personality disorder symptoms will be measured using Zanarini Rating Scale for Borderline Personality Disorder (ZAN-BPD) - self-report version. Scores range from 0-36; higher scores indicate greater severity of borderline personality disorder symptoms
Change in clinician-rated clinical severity | 44 weeks (baseline, post-treatment/waitlist, 6 month follow-up)
  Clinical severity will be measured using the Diagnostic Interview for Anxiety, Mood, and Obsessive Compulsive and Related Neuropsychiatric Disorders (DIAMOND) dimensional clinician ratings. Scores range from 1-7; higher scores indicate greater severity.
Change in Anxiety Symptoms | 12 weeks (baseline, week 1, week, 2, week, 3.....week 12)
  Anxiety symptoms will be measured using the Overall Anxiety Severity and Interference Scale (OASIS). This is a self-report measure in which scores range from 0-20; higher scores indicate more severe anxiety symptoms.
Change in Depressive Symptoms | 12 weeks (baseline, week 1, week, 2, week, 3.....week 12)
  Depressive symptoms will be measured using the Overall Depression Severity and Interference Scale (ODSIS). This is a self-report measure in which scores range from 0-20; higher scores indicate more severe anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Sauer-Zavala, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sauer-Zavala S, Southward MW, Fruhbauerova M, Semcho SA, Stumpp NE, Hood CO, Smith M, Elhusseini S, Cravens L. BPD compass: A randomized controlled trial of a short-term, personality-based treatment for borderline personality disorder. Personal Disord. 2023 Sep;14(5):534-544. doi: 10.1037/per0000612. Epub 2023 Jan 2. PMID 36595435